CLINICAL TRIAL: NCT00541801
Title: Acoustic Cardiographic Assessment of Heart Function in Comparison to Doppler-echocardiography in Patients With Cytostatic Therapies
Brief Title: Acoustic Cardiographic Assessment of Heart Function in Comparison to Doppler-echocardiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Collaborators: Inovise Medical (Industry)
Responsible Party: Paul Erne, Kantonsspital Luzern
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Audicor-Oncology
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Heart Failure, Congestive; Antineoplastic Agents
MeSH Terms: conditions — Heart Failure | interventions — Echocardiography, Doppler

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Doppler-echocardiography and acoustic cardiography — Patients receive a Doppler-echocardiography and an acoustic cardiography

SUMMARY:
In this study, the investigators sought to determine whether an acoustic cardiographic assessment of heart function is equivalent to Doppler-echocardiography in patients who are treated with cardio-toxic cytostatic agents.

DETAILED DESCRIPTION:
Patients receiving cardio-toxic cytostatic agents are examined by Doppler-echocardiography and acoustic cardiography before, during, and after the cytostatic treatment. Doppler-echocardiography measures ejection fraction, TDI, speckle tracking, and further parameters. Acoustic cardiography (Audicor, Inovise Medical Inc., Portland, USA) simultaneously integrates heart sounds and single-channel electrocardiography input to generate multiple parameters that correlate to established hemodynamic measures. Heart function as assessed by Doppler-echocardiography is then compared to the heart function as assessed by Audicor ECG.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant disease with scheduled anthracycline and trastuzumab therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Changes of echocardiographic parameters and changes of electromechanical activation time (EMAT)and development of third heart sound as indicators of congestive heart failure | Repeated measurements over a year

SECONDARY OUTCOMES:
Development of clinically overt congestive heart failure | One year

CONTACTS AND LOCATIONS:
Overall Officials: Paul Erne, MD, Study Chair — Luzerner Kantonsspital
Locations (1):
- Kantonsspital Luzern, Department of Cardiology, Lucerne, Canton of Lucerne, Switzerland